CLINICAL TRIAL: NCT00884897
Title: Oxytocin and Social Cognition in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, MPRC, Deanna L. Kelly, Pharm.D., BCPP, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00041024; P50MH082999 (NIH)
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Social Cognition; Social Anxiety; Emotional Intelligence
Keywords: Social Cognition; Schizophrenia; Oxytocin
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): We will purchase OT from PharmaWorld, an international pharmacy located in Switzerland; the preparation of intranasal OT is manufactured by Novartis and sold under the trade name: Syntocinon. We have obtained an IND (number 78,246) for Syntocinon (intranasal oxytocin) manufactured by Novartis.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): We will be purchasing oxytocin placebo nasal spray through LABOSWISS located in Davos, Switzerland and distributed through PharmaWorld. LABOSWISS will manufacture the matching the placebo under GDP guidelines. The placebo will be in every way identical to the oxytocin formulation but will not contain OT.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Oxytocin given as 20 IU BID
  Arms: Oxytocin
Drug: Placebo — Placebo given as 20 IU BID
  Arms: Placebo

SUMMARY:
Objective: Social Cognition and Emotional Intelligence have been shown to be deficient in patients with schizophrenia and these are not remediated by antipsychotic medications or psychosocial interventions. Social cognition is associated with functional outcome, an important step in striving for recovery in this population. The hormone and neurotransmitter, oxytocin, which has been associated with social bonding and trust has been shown to improve measures of some aspects of social cognition in humans. The study will assess the effect of acute administration of intranasal oxytocin on measures of social cognition and functioning as well as on emotional intelligence and symptoms.

Study population: The study population will include patients with a DSM-IV diagnosis of schizophrenia or schizoaffective disorder who have been on a stable medication regimen for 6 weeks. We will enroll a total of 30 subjects (N=15 placebo and N=15 oxytocin groups).

Experimental design and methods: After a one week lead in phase, participants will undergo 3 weeks of oxytocin (20 IU BID) or placebo administration (double blind) in addition to their existing medication regimen. Outcome measures will be administered during the lead in phase, and at the end of the study drug administration phase (under the acute effect of OT). The primary outcome measure will be the Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) and the Maryland Assessment of Social Competence (MASC). Secondary measures include rating from the domains of social cognition (emotion perception, attributional style, theory of mind and social perception), symptom rating and measures of social anxiety and quality of life. Side effects and symptoms will be measured weekly.

ELIGIBILITY:
Inclusion criteria:

All participants must:

1. Be between age 18 and 55.
2. Meet DSM-IV criteria for Schizophrenia or Schizoaffective Disorder.
3. Treated with a stabilized antipsychotic regimen (i.e., have had no change in antipsychotic medication in the previous six weeks and no change in dose for the past 30 days).

Exclusion criteria:

Participants will be excluded if they have evidence of:

1. DSM-IV criteria for substance dependence in the last 6 months or DSM-IV criteria for abuse in the past 30 days.
2. Cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires. This is defined an as a score of less than 10 on the Evaluation to Sign Consent (ESC) and judged by the treating clinician.
3. Medical illness that in the view of the investigators would compromise participation in research.
4. History of polydipsia and/or hyponatremia
5. Clinically significant endocrine disorders, as judged by the PI. Abnormalities in prolactin levels and thyroid function tests associated with the use of dopamine antagonist medications will not be exclusionary.
6. Pregnancy, planning to become pregnant, or breastfeeding. In addition, women of childbearing age are required to use an effective form of birth control for the duration of the study. Effective forms of birth control include:

   * hormonal contraceptives (birth control pills, injectable hormones, vaginal ring hormones),
   * surgical sterility (tubal ligation or hysterectomy)
   * IUD
   * Diaphragm with spermicide
   * Condom with spermicide
   * Abstinence
7. Use of any drugs (prostaglandins, vasoconstricting agents or anesthetic medications, for example) that may interact with oxytocin. Justification: Avoidance of adverse interaction with oxytocin. Assessment tool(s): Clinical interview and toxicology screen
8. History of hypersensitivity to oxytocin or vehicle, i.e. propyl parahydroxybenzoate, methyl parahydroxybenzoate, chlorobutanol hemihydrate. Assessment tool: clinical interview
9. Presence of or history of clinically significant allergic rhinitis as assessed by the PI, M.D., or Nurse. Justification: Inflammation of nasal mucosa could interfere with mucosal absorption of intranasally administered OT. Current rhinitis from an upper respiratory infection should be resolved prior to enrollment in study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, Pharm.D, BCPP, Principal Investigator — University of Maryland, College Park; Mary Lee, MD, Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- Maryland Psychiatric Research Center (MPRC) Outpatient Research Program (ORP); the MPRC Treatment Research Program (TRP), Catonsville, Maryland, United States

REFERENCES:
- [Derived] Lee MR, Wehring HJ, McMahon RP, Liu F, Linthicum J, Verbalis JG, Buchanan RW, Strauss GP, Rubin LH, Kelly DL. Relationship of plasma oxytocin levels to baseline symptoms and symptom changes during three weeks of daily oxytocin administration in people with schizophrenia. Schizophr Res. 2016 Apr;172(1-3):165-8. doi: 10.1016/j.schres.2016.02.014. Epub 2016 Feb 12. PMID 26879587
- [Derived] Lee MR, Wehring HJ, McMahon RP, Linthicum J, Cascella N, Liu F, Bellack A, Buchanan RW, Strauss GP, Contoreggi C, Kelly DL. Effects of adjunctive intranasal oxytocin on olfactory identification and clinical symptoms in schizophrenia: results from a randomized double blind placebo controlled pilot study. Schizophr Res. 2013 Apr;145(1-3):110-5. doi: 10.1016/j.schres.2013.01.001. Epub 2013 Feb 13. PMID 23415472

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 13 | 15
Completed | 13 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline participants are participants that were randomized to one of the two treatment groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.74 (11.74) | 35.07 (8.21) | 39.6 (11.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 15 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: To Determine Whether Exogenous OT Enhances Emotional Intelligence and Improves Performance on Measures of Social Cognition for Schizophrenia or Schizoaffective Patients
Description: Mayer-Salovay Caruso Emotional Intelligence Test (Mayer et al., 2002; MSCEIT) This is a self report instrument that consists of 141 items and 8 ability subscales, which assess four components (branches) of emotion processing: identifying emotions, using emotions, understanding emotions, and managing emotions. For this study we will focus on the managing emotions and understanding emotions components. There are 29 total items assessed with a total score ranging from 5-145. The higher the score the better the outcome.
Time Frame: participants are assessed at baseline and end point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 13 | 15
units on a scale
  Understanding Emotions (Baseline) | 82.2 (12.4) | 77.9 (9.8)
  Understanding Emotions (Endpoint) | 76.7 (9.2) | 84.3 (10.4)
  Managing Emotions (Baseline) | 87.1 (10.0) | 77.9 (9.8)
  Managing Emotions (Endpoint) | 76.7 (9.2) | 84.3 (10.4)

2. Secondary Outcome: To Determine Whether OT Improves Measures of Social Anxiety.
Description: To determine whether OT improves measures of social anxiety as measured by the Social Interaction Anxiety Scale. This assessment has 20 items scored 0-4 for a total minimum score of 0 and maximum score of 80. The lower the score the better the outcome.
Time Frame: Outcomes are compared between Baseline and endpoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 13 | 15
units on a scale
  Baseline | 30.1 (14.4) | 33.9 (17.8)
  4 Weeks (Endpoint) | 26.4 (12.0) | 26.1 (14.2)

ADVERSE EVENTS:
Arm/Group | Oxytocin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 9/13 | 10/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=13) | Placebo (N=15)
Vomiting (Gastrointestinal disorders) | 1 | 0 (0)
Abdominal pain (General disorders) | 3 | 3
Anorexia (General disorders) | 0 | 1
Constipation (General disorders) | 1 | 1
Diarrhea (General disorders) | 1 | 2
Dizziness (General disorders) | 1 | 2
Dry mouth (General disorders) | 1 | 3
Fever (General disorders) | 1 | 0
Headache (General disorders) | 1 | 4
Insomnia (General disorders) | 3 | 4
Malaise (General disorders) | 2 | 1
Nausea (General disorders) | 4 | 1
Restlessness (General disorders) | 4 | 4
Salivation (General disorders) | 3 | 1
Sedation (General disorders) | 3 | 1
Sore throat (General disorders) | 0 | 2
Stiffness (General disorders) | 2 | 1
Tinnitus (General disorders) | 0 | 2
Tremor (General disorders) | 2 | 2
Urticaria (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No